CLINICAL TRIAL: NCT05866380
Title: Early Identification of Heart Failure in Diabetes With Known Cardiovascular Risk or Established Cardiovascular Disease in A Large-scale Asian Diabetic Population: A Multi-center Cohort Study
Brief Title: Early Identification of Heart Failure in a High-Risk Diabetic Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung-Lieh Hung, Doctor, Mackay Memorial Hospital
Other Study IDs: 20MMHIS365e
Record Dates: First submitted 2023-05-08; First posted 2023-05-19 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Type2diabetes
Keywords: Type2diabetes; Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: heart failure risk factors — observational study with diabetes patient with heart failure risk factors

SUMMARY:
Type 2 diabetes is an important co-morbid condition strongly associated with the risk of developing heart failure (HF). Risk scores such as the WATCH-DM score that predict the occurrence of HF among diabetes patients are largely based on data collected from white ethnicities. Here, the investigators sought to investigate surrogate markers for predicting HF among type 2 diabetes patients of Asian ethnicities.

DETAILED DESCRIPTION:
Patients with type 2 diabetes (T2D) suffer from diverse complications, including atherosclerotic cardiovascular disease (ASCVD), diabetic cardiomyopathy and heart failure (HF), which accounts for a substantial burden of death and disability worldwide. Epidemiological studies have pointed out the projected global diabetes trends with estimated 642 million by 2040. On the other hand, patients with HF are accompanied by high burden of T2D, which in turn exacerbate grave prognosis of HF. Despite the observed benefits in controlling risk factors of hypertension, ...etc. in preventing incident HF, efforts has lead to little effect from strict sugar control in diabetic patients.

Recent cardiovascular outcomes trials (CVOTs) have shown substantial improvement on cardiovascular protective effects and end-points with novel SGLT2 inhibitors, particularly in HF, yet data regarding the exact clinical characteristics and risk stratification in diabetes subjects that interventions may help remained largely unexplored. To date, several baseline clinical information along with biomarker N-terminal pro-brain natriuretic peptide (NT-proBNP) have shown to be predictors of HF. According to WATCH-DM sub-study based on The Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial, a variety of clinical variables, including age, gender, body size, blood pressure, dys-glycemic indices and lipid profiles haven shown to identify the clinical risks for HF in T2D patients. Beyond clinical risk factors, biomarkers of NT-proBNP, a sensitive serum marker for cardiac damage and pre-clinical myocardial dysfunction, has also shown novelty in identifying diabetic subjects with subclinical cardiac dysfunction or with higher HF risk starting from relatively lower clinical cut-offs (NTproBNP≧50 pg/mL) that may benefit from SGLT2i treatment.

This trial is a multi-center clinical study in Mackay Memorial Hospital, National Taiwan University Hospital and Far Eastern Memorial Hospital. A total 5000 adult T2D patients will be prospectively enrolled from outpatient clinics (1500-3500 patients each center). 5000 - 10000 retrospective medical record reviews (3000 - 7000 each center) for baseline characteristics and general biochemical examination results collection ( including blood sugar, glycated hemoglobin, lipid profile, liver function, renal function and microalbuminuria), EKG. WATCH-DM score collection and heart function related biomarkers test including NTproBNP will be arranged.

Through the value of biomarker detection, high-risk type 2 diabetes patients who have not previously caused heart disease can be identified, and the epidemiology of high-risk Asian type 2 diabetes with preclinical HF will be elucidated by large-scale cohort research.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes T2DM for at least six months;
* ≥ 20 years of age, men or women;
* Patients who had either established cardiovascular disease or additional cardiovascular risk factors;
* Free at baseline of diagnosed HF, while patients might be stage A-B HF based on ACC/AHA Heart Failure Classification, with baseline clinical information and NTproBNP data available;
* Baseline patient-level clinical data available.

Exclusion Criteria:

* eGFR <30ml/min/1.73m2;
* Known HF hospitalization history;
* Known impaired LV systolic function (LVEF<40%) by any imaging modality;
* Any terminal disease other than diabetes lowering the patient's life expectancy to less than two years;
* Pregnant women.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM patients, ethnic Asians, with established cardiovascular diseases or additional cardiovascular risk factors
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | From date of recruitment until the date of first documented progression, with the minimum of 12 months of follow-up.
  Major adverse cardiovascular events defined as a composite of hospitalization for heart failure, death from cardiovascular causes and nonfatal myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Lieh Hung, MD.PhD, Principal Investigator — MackayMemorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No